CLINICAL TRIAL: NCT01180374
Title: Cannabidiol Modulation of ∆-9-THC's Psychotomimetic Effects in Healthy Humans
Brief Title: The Effects of Cannabidiol and ∆-9-THC in Humans
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Mohini Ranganathan, Principal Investigator, Yale University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1001006240
Record Dates: First submitted 2010-08-10; First posted 2010-08-12 (Estimated); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Healthy
Keywords: Cannabis; Marijuana; Cannabidiol; CBD; THC; Psychotic Disorders
MeSH Terms: conditions — Marijuana Abuse; Psychotic Disorders | interventions — Cannabidiol; Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Active Canabidiol and Active Delta-9-THC (Experimental)
  Interventions: Drug: Cannabidiol; Drug: Delta-9-THC
- Placebo and Active Delta-9-THC (Placebo Comparator)
  Interventions: Drug: Delta-9-THC; Drug: Placebo
- Active Cannabidiol and Placebo (Experimental)
  Interventions: Drug: Cannabidiol; Drug: Placebo
- Placebo and Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol — Active Cannabidiol 5mg.
  Arms: Active Canabidiol and Active Delta-9-THC; Active Cannabidiol and Placebo
Drug: Delta-9-THC — Active Delta-9-THC (0.035mg/Kg) given intravenously over 20 minutes. The dose of THC that you may receive is a small dose and is roughly equivalent to smoking approximately one half to one whole marijuana cigarette, or "joint".
  Arms: Active Canabidiol and Active Delta-9-THC; Placebo and Active Delta-9-THC
Drug: Placebo — Placebo (about a quarter spoon of alcohol with no CBD).
  Arms: Placebo and Active Delta-9-THC; Placebo and Placebo
Drug: Placebo — Placebo (about a quarter spoon of alcohol with no THC) given intravenously over 20 minutes.
  Arms: Active Cannabidiol and Placebo; Placebo and Placebo

SUMMARY:
Cannabis is the most commonly used illicit substance in the US and herbal cannabis consists of a number of cannabinoids including Δ-9 THC and CBD. This study will characterize the interactive effects of the two major components of cannabis i.e. Δ-9-THC and CBD.

ELIGIBILITY:
Inclusion Criteria:

* Exposed to Cannabis at least once in lifetime

Exclusion Criteria:

* Cannabis Naive

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2010-02-01 (Actual); Primary Completion 2014-10-06 (Actual); Study Completion 2014-10-06 (Actual)

PRIMARY OUTCOMES:
Behavioral Measures | Baseline, +15, +80, +240
  Subjective effects, perceptual alterations, and cognitive effects will be assessed using visual analog scales, Positive and Negative Symptom Subscale (PANSS), Clinician Administered Dissociative States Scale (CADSS), Psychotomimetic States Inventory (PSI) and a neuro cognitive battery.

CONTACTS AND LOCATIONS:
Overall Officials: Mohini Ranganathan, M.D, Principal Investigator — Yale University Medical School
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

REFERENCES:
- [Derived] Ganesh S, Cortes-Briones J, Schnakenberg Martin AM, Skosnik PD, D'Souza DC, Ranganathan M. Delta-9-Tetrahydrocannabinol, Cannabidiol, and Acute Psychotomimetic States: A Balancing Act of the Principal Phyto-Cannabinoids on Human Brain and Behavior. Cannabis Cannabinoid Res. 2023 Oct;8(5):846-856. doi: 10.1089/can.2021.0166. Epub 2022 Mar 18. PMID 35319274